CLINICAL TRIAL: NCT03820856
Title: Therapeutic Effects of Acupuncture Plus Fire Needle Versus Acupuncture on Lateral Epicondylitis: A Randomized Case-control Pilot Study
Brief Title: Acupuncture Plus Fire Needle and Acupuncture on Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 98-3818A3
Record Dates: First submitted 2019-01-24; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2010-03

CONDITIONS: Lateral Epicondylitis; Tennis Elbow; Acupuncture
Keywords: Lateral Epicondylitis; Tennis Elbow; Acupuncture; Fire needle
MeSH Terms: conditions — Tennis Elbow | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture plus fire needle group (Experimental)
  Interventions: Procedure: acupuncture plus fire needle therapy
- acupuncture group (Active Comparator)
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture plus fire needle therapy — The protocol used in this group was the same as that used in the acupuncture alone group except that fire needle therapy was added. The treatments were administered twice weekly for 6 weeks. Fire needle therapy was performed as follows: an acupuncture needle made of tungsten was heated until red-hot over a lighter and then inserted into the two Ah shi points (the tender points on the common extensor tendon, specifically extensor carpi radialis). The red-hot needle was inserted rapidly into the Ah shi point (approximately 5-8 fen deep, 1 cun = 10 fen) for approximately half a second and then removed. Pressure was then applied to the needle hole using a sterilized dry cotton ball.
  Arms: acupuncture plus fire needle group
Procedure: acupuncture — We selected acupoints that have often been recommended for the treatment of lateral epicondylitis. Triple needling was performed at the Ah shi point, i.e., the 1-2-cm area encompassing the most painful spot on the humeral epicondyle. We also manipulated acupuncture needles in the following areas: LI10 (Shousanli), LI11 (Quchi), LI12 (Zhouliao) and LU5 (Chize). The treatments were administered twice weekly for 6 weeks.
  Arms: acupuncture group

SUMMARY:
The aim of this study was to investigate whether or not the outcomes of acupuncture used in combination with fire needle treatment are better than those of acupuncture alone in patients with lateral epicondylitis.

The primary outcome was the visual analog scale pain score for the previous 24 hours and the secondary outcomes were the maximum grip strength, Patient-rated Forearm Evaluation Questionnaire score, and Medical Outcomes Study 36-Item Short-form Health Survey score. The values at baseline (pretreatment), at the end of treatment, and at three months after treatment were used to assess the short-term and intermediate-term effects of treatment.

DETAILED DESCRIPTION:
Lateral epicondylitis (LE) is the most common diagnosis in patients with elbow pain.

Although many management strategies have been used in patients with LE, including pain-relieving drugs, corticosteroid injections, physiotherapy, elbow supports, shock-wave therapy, platelet-rich plasma injections, and surgery, the optimal treatment is still unclear. When conservative treatments are unsuccessful or not accessible because for cost reasons, an increasing number of patients consider complementary medicine, particularly acupuncture.

In a systematic review by Trinh et al., acupuncture was found to relieve the pain of LE effectively but its long-term efficacy could not be established. Another technique commonly used to treat chronic pain in patients with LE is fire needle therapy, which combines acupuncture and moxibustion. A case report demonstrated a significant short-term effect of fire needle therapy in a patient with LE. Moreover, it has been shown that a combination of rehabilitation and fire needle therapy is effective for at least 4 weeks in patients with LE. However, although the early case report demonstrated effects lasting for 4 months, there was insufficient evidence for the intermediate-term or long-term therapeutic effects of acupuncture or fire needle therapy in terms of reducing the pain associated with LE.

The aim of this study was to investigate whether or not the outcomes of acupuncture used in combination with fire needle treatment are better than those of acupuncture alone in patients with LE.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were selected for inclusion if two or more of the following criteria were noted on the physical examination form: pain over the lateral aspect of the elbow; pain on palpation over the lateral epicondyle or the associated myotendinous junction of the common extensor tendon; pain on hand gripping; and pain with either resisted static contraction or stretching of the wrist extensor muscles.
2. symptoms have persisted for at least 2 months
3. symptoms are unilateral

Exclusion Criteria:

1. signs and symptoms suggesting a cause other than overuse (e.g., cervical radiculopathy)
2. osteoarthritis of the elbow joints
3. pathologic, neurologic, and/or vascular findings in the arms
4. arthritis (local/generalized polyarthritis)
5. radiohumeral bursitis
6. ligamentous sprain
7. bilateral tennis elbow
8. painful shoulder
9. surgery or dislocation of the elbow
10. coagulopathy
11. pregnancy
12. infection
13. malignancy
14. Patients who had been treated with other therapies or drugs for lateral epicondylitis in the 2 weeks before the start of the trial, those who had received corticosteroid injections in the previous 6 months, and those who had received acupuncture and fire needle therapy for lateral epicondylitis were also excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-08-05 (Actual); Primary Completion 2011-03-18 (Actual); Study Completion 2011-03-18 (Actual)

PRIMARY OUTCOMES:
changes in severity of elbow pain (VAS score) | baseline, 6 weeks, 18 weeks
  The severity of the patient's elbow pain was evaluated using a 10-point VAS (0, no pain; 10, most severe pain imaginable) at rest, during motion, and on exertion.

SECONDARY OUTCOMES:
changes in maximum grip strength | baseline, 6 weeks, 18 weeks
  The patient is required to stand with his or her arm alongside the body with the forearm pronated and the elbow extended while holding the dynamometer. The patient is then instructed to squeeze once with maximum pressure, and the measurement is recorded. The maximum grip strength is measured three times with a 30-second rest interval between each measurement.
changes in Patient-rated Forearm Evaluation Questionnaire score | baseline, 6 weeks, 18 weeks
  The Patient-rated Forearm Evaluation Questionnaire is useful for assessment of the outcome of treatment for lateral epicondylitis. The Patient-rated Forearm Evaluation Questionnaire is divided into two sections, ie., pain and function at the elbow.
changes in Medical Outcomes Study 36-Item Short-form Health Survey score | baseline, 6 weeks, 18 weeks
  Quality of life was assessed using the Study 36-Item Short-form Health Survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan